CLINICAL TRIAL: NCT05702788
Title: A Multicenter, Randomized, Double-blind, Placebo-parallel Controlled Study to Evaluate the Efficacy and Safety of Jaktinib Hydrochloride Tablets in Participants Receiving the Best Available Treatment for Severe Novel Coronavirus Pneumonia
Brief Title: Efficacy and Safety of Jaktinib in Participants With Severe Novel Coronavirus Pneumonia(COVID-19)
Acronym: COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor R&D Strategy Adjustment
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAK032
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jaktinib 75mg BID (Experimental): Jaktinib 75mg BID
  Interventions: Drug: Jaktinib hydrochloride tablets
- Jaktinib 100mg BID (Experimental): Jaktinib 100mg BID
  Interventions: Drug: Jaktinib hydrochloride tablets
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Jaktinib hydrochloride tablets — 75mg of Jaktinib administered orally Twice daily(BID) with best available treatment.
  Arms: Jaktinib 75mg BID
Drug: Jaktinib hydrochloride tablets — 100mg of Jaktinib administered orally Twice daily(BID) with best available treatment.
  Arms: Jaktinib 100mg BID
Other: Placebo — Placebo (given as two placebo tablets) administered orally BID with best available treatment.
  Arms: Placebo

SUMMARY:
This study adopts a randomized, double-blind, placebo parallel control design, and is expected to include 168 eligible patients with severe novel coronavirus pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, male or female;
* The Participants was diagnosed with novel coronavirus pneumonia;
* It meets the heavy-duty standards of the new coronavirus pneumonia diagnosis and treatment protocol (version 9).
* Participants who voluntarily sign informed consent.
* The National Institute of Allergy and Infectious Diseases Sequential Scale (NIAID-0S) score is 5 or 6;

Exclusion Criteria:

* Participants who cannot take orally, or are suspected to be allergic to Jaktinib, similar drugs or their excipients, or have severe gastrointestinal dysfunction that affects drug absorption;
* Participants who have received the following treatments within the specified time window before randomization:

  1. Participants have received Janus kinase (JAK) inhibitor, interleukin 6 (IL-6) inhibitor, IL-1 inhibitor, tumor necrosis factor (TNF) inhibitor, T cell or B cell depletion agent, interferon and other immunosuppressive drugs within the first two weeks of randomization, except glucocorticoid;
  2. Systematically used CYP 3A4 potent inhibitor or potent inducer in the first five drug half lives at random;
* Immune deficiency;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
The proportion of Participants who develop death or respiratory failure. | 28 days after randomization
  Respiratory failure is defined as Participants who on invasive mechanical ventilation or Extracorporeal Membrane Oxygenation(ECMO) or on non-invasive ventilation or high-flow oxygen devices.

SECONDARY OUTCOMES:
The proportion of Participants who develop death or respiratory failure. | 14 days after randomization
  Respiratory failure is defined as Participants who on invasive mechanical ventilation or ECMO or on non-invasive ventilation or high-flow oxygen devices.

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, Principal Investigator — The Third People Hospital of Shenzhen

IPD SHARING:
Plan to Share IPD: No